CLINICAL TRIAL: NCT00880412
Title: A Pilot, Randomized, Double-blind, Placebo-controlled, Parallel Group, Multicentre, Phase IIA Study to Determine the Clinical Safety/Tolerability and Exploratory Efficacy of EHT 0202 (40 and 80 mg Bid) as Adjunctive Therapy to Acetylcholinesterase Inhibitor Over a 3-month Period in Ambulatory Patients Suffering From Mild to Moderate Alzheimer's Disease (EHT 0202/002 Protocol)
Brief Title: A Study to Determine the Clinical Safety/Tolerability and Exploratory Efficacy of EHT 0202 as Adjunctive Therapy to Acetylcholinesterase Inhibitor in Mild to Moderate Alzheimer's Disease
Acronym: EHT0202/002
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Exonhit (Industry)
Responsible Party: Professor Bruno Vellas, MD, University of Toulouse - Purpan - Casselardit Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EHT0202/002
Record Dates: First submitted 2009-04-10; First posted 2009-04-13 (Estimated); Last update posted 2009-09-21 (Estimated); Status verified 2009-09

CONDITIONS: Alzheimer's Disease
Keywords: safety; efficacy; Alzheimer's disease; treatment; phase II; study; cholinesterase inhibitor
MeSH Terms: conditions — Alzheimer Disease | interventions — Etazolate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- EHT 0202 40 mg bid (Experimental): study treatment is given in addition to one acetylcholinesterase inhibitor (galantamine, rivastigmine or donepezil)
  Interventions: Drug: EHT 0202 etazolate
- EHT 0202 80 mg bid (Experimental): study treatment is given in addition to one acetylcholinesterase inhibitor (galantamine, rivastigmine or donepezil)
  Interventions: Drug: EHT 0202 etazolate
- placebo bid (Placebo Comparator): study treatment is given in addition to one acetylcholinesterase inhibitor (galantamine, rivastigmine or donepezil)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EHT 0202 etazolate — In each arm, 2 capsules of study treatment (capsules of EHT0202 40mg and/or placebo) are taken twice a day during breakfast and dinner over a 3-month treatment period. There is non treatment adjustment.
  Other Names: EHT 0202; etazolate
  Arms: EHT 0202 40 mg bid; EHT 0202 80 mg bid
Drug: Placebo — In each arm, 2 capsules of study treatment (capsules of EHT0202 40mg and/or placebo) are taken twice a day during breakfast and dinner over a 3-month treatment period. There is non treatment adjustment.
  Arms: placebo bid

SUMMARY:
The objective of this 3-month study is to assess the safety and efficacy of EHT 0202 in addition to acetylcholinesterase inhibitor in patients suffering from Alzheimer's Disease.

DETAILED DESCRIPTION:
The aim of this pilot study is to assess the safety and tolerability profile of 2 doses of EHT 0202 (40 mg and 80 mg b.i.d) versus placebo in addition to a treatment with acetylcholinesterase inhibitor and its exploratory efficacy on cognition, behavior, activities of daily living, caregiver's burden and patient's global assessment, during a 3-month treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory male or female patient, aged 60-90 years old included at screening, and living at home.
* Patient having a clinical diagnosis of probable AD according to National Institute of Neurological and Communicative Disorders and Stroke/Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria.
* Mild to moderate AD with a MMSE total score ≥ 12 and ≤ 24 at screening.
* Written informed consent obtained from the patient or, if appropriate, from legal representative according to local laws and regulations. The caregiver will also have to sign a specific informed consent form regarding his/her participation in the study.
* Patient treated for AD treatment with one AChEI (donepezil, galantamine, or rivastigmine), according to the recommended posology mentioned in the summary of product characteristics, for at least 3 months and with a stable dose for at least 2 months prior to screening. The dose should be kept unchanged throughout the study duration.
* Patient with a cerebral CT-scan or cerebral MRI compatible with AD diagnosis, with no brain lesions that may be related to another diagnosis and that could be responsible for the current patient's condition (ex, but not limited to, non-AD dementia, brain injury, brain tumour, stroke, normal pressure hydrocephalus,…). A cerebral CT-scan or cerebral MRI has to be performed and results have to be available prior patient's randomization if the results of the brain imagery performed to settle the AD diagnosis are not available in the patient's file. Brain imaging has also to be performed if considered necessary by the investigator, such as in case of emerging neurological symptoms or in case of worsening of existing neurological symptoms.
* Neurological exam without any particularities or without any specific focal signs likely to be related to other conditions than AD.
* No contra-indication to AChEI treatment and absence of significant adverse events considered to be related to AChEI treatment at screening and randomisation.
* Patient and patient's caregiver able to comply with study procedures, notably regarding the drug intake at the end of the meal which has to be supervised by the caregiver or another competent person.

Exclusion Criteria:

* Diagnosis of vascular dementia according to NINDS-AIREN criteria, or other non-AD dementia, or CNS pathology (including but not limited to brain injury, brain tumour, stroke, normal pressure hydrocephalus, Parkinson's disease, epilepsy,multiple sclerosis,…) that may be responsible for dementia.
* Clinically significant pathology and/or uncontrolled condition, including but not limited to cancer, infectious (like AIDS), gastro-intestinal, hepatic, renal, respiratory, endocrine(like diabetes mellitus, thyroiditis) pathology.
* History or current clinically significant psychiatric pathology (including but not limited to psychotic disorders, bipolar disorder, personality disorders) that may interfere with study assessments.
* Current major depressive disorder, either treated or not, associated with clinically significant symptoms.
* Low blood level of vitamin B12, TSH levels out of normal range at screening.
* Current forbidden medication intake or intake within 2 weeks prior to screening.
* Recent history (within the past year prior to inclusion) or current cardiovascular pathology and/or symptoms considered as clinically significant, including but not limited to angina pectoris, uncontrolled arrhythmia, significant ECG abnormalities. Lifetime history of heart failure, myocardial infarction, severe and/or uncontrolled angina pectoris,and/or ventricular arrhythmia disqualifies the patient.
* History or presence of clinically conditions that may interfere with product metabolism or with study assessments.
* Systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 90 mmHg at screening and/or randomisation.
* QTc interval (Bazett's correction) ≥ 430 msec for male and ≥ 450 msec for female at screening.
* Laboratory values (biochemistry, haematology, urinalysis) considered as clinically significant and/or that may interfere with study assessments, according to the investigator.
* ALAT, ASAT, ALP > 2.5 times the upper normal limit (UNL), total bilirubin > 1.5 UNL or history of significant liver pathology including hepatitis caused by drugs, HBV, HCV.
* BUN, creatinin > 1.5 UNL.
* Current or recent history of drug or alcohol abuse or dependence.
* Patient not registered at "Sécurité Sociale".
* Participation in another study within 1 month prior to screening and during the whole duration of the study.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2008-04; Primary Completion 2009-06 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
incidence/frequency and severity of adverse events, relation to treatment start and drug exposure, drop-out rate, including reason for withdrawal, clinical examination, change from screening of biological safety parameters, vital signs, ECG and weight. | all study visits

SECONDARY OUTCOMES:
Assessment of cognition (ADAS-Cog, Neuropsychological Test Battery, MMSE), patient's global functioning (CDR-SB,CGI), patient's behaviour (NPI), daily living activities (ADCS-ADL) and caregiver's burden. Population PK of EHT 0202 and PK/PD profile. | at the end of the 3-month study treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Vellas, MD, Principal Investigator — Casselardit Hospital - University of Toulouse
Locations (22):
- France (22):
  - Hôpital Privé Les Magnolias, Ballainvilliers
  - Cabinet Médical, Bergerac
  - Fleyriat Hospital, Bourg-en-Bresse
  - Cabinet Médical, Dijon
  - Charles Foix Hospital, Ivry-sur-Seine
  - Cabinet Médical, La Seyne-sur-Mer
  - Roger Salengro Hospital, Lille
  - Dupuytren Hospital, Limoges
  - Clinique Léopold Bellan, Magnanville
  - Cabinet Médical, Montpellier
  - Cabinet Médical 2, Montpellier
  - CHU Nantes Hôpital Laennec, Nantes
  - Cabinet Médical 2, Nice
  - Cabinet Médical, Nice
  - CHU Cochin Broca, Paris
  - Cabinet Médical, Rambouillet
  - CHU Rennes, Rennes
  - Cabinet Médical, Rodez
  - Cabinet Médical, Rueil-Malmaison
  - Cabinet Médical, Saint-Brieuc
  - Cabinet Médical, Toulon
  - Purpan-Casselardit Hospital - University of Toulouse, Toulouse